CLINICAL TRIAL: NCT06793293
Title: Effect of High Level Laser Therapy on Postoperative Cesarean Section Incisional Pain
Brief Title: Postoperative in Cesarean Section, the Women Suffering from Pain Due to Wound "incisional Pain", High Level Laser One of Most Effective Methods That Promoting Healing and Decrease Pain so It Will Effective If Use in Decreasing Pain of Cesarian Section
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ibrahim Awad Shweal, Teacher assistance at faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.Rec/012/005570
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cesarean Section Pain
Keywords: cesarean section pain; High power laser; decreasing pain; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: High power level laser used after cesarian section to decrease pain for 3 sessions first, second and third day.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High level laser (Experimental): It will be consisted of twenty-five postoperative cesarean section women and will be treated by medical treatment (Non-steroidal anti- inflammatory drugs and antibiotics) in addition to High level laser for 5 minutes on days 1 st , 2 nd , and 3 rd , after cesarean section (3 sessions)
  Interventions: Device: High level laser
- (Non-steroidal anti- inflammatory drugs and antibiotics) (Active Comparator): It will be consisted of twenty-five postoperative cesarean section women and will be treated by medical treatment (Non-steroidal anti- inflammatory drugs and antibiotics) only.
  Interventions: Drug: Non-steroidal anti- inflammatory drugs and antibiotics

INTERVENTIONS:
Device: High level laser — It will be consisted of twenty-five postoperative cesarean section women and will be treated by medical treatment (Non-steroidal anti- inflammatory drugs and antibiotics) in addition to High level laser for 5 minutes on days 1 st , 2 nd , and 3 rd , after cesarean section (3 sessions)
  Other Names: High power laser
  Arms: High level laser
Drug: Non-steroidal anti- inflammatory drugs and antibiotics — It will be consisted of twenty-five postoperative cesarean section women and will be treated by medical treatment (Non-steroidal anti- inflammatory drugs and antibiotics) only.
  Arms: (Non-steroidal anti- inflammatory drugs and antibiotics)

SUMMARY:
High power laser is safe and effective methods, it's uses increasing one day after day in decreasing pain and promoting healing so its use in postoperative cesarian section will help mothers to overcome pain and return to ADLs faster

ELIGIBILITY:
Inclusion Criteria:

* Their ages will be ranged from 20-40 years. 2. Their BMI will be less than 30 Kg\m 2 3. Patients with lower segment cesarean section (Poursalehan et al., 2018 & de Holanda et al., 2020).

Exclusion Criteria:

* 1. Patients with upper segment cesarean section. 2. Diabetic patient. 3. Patient with malignancy, benign tumors with the possibility to become malignant. 4. Infection of the skin (Poursalehan et al., 2018).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS): | third day
  It will be used to assess the severity of low back pain in women from both groups A and B before and after treatment. The scoring ranges from 1, indicating the least pain and discomfort, to 10, representing the most severe pain and discomfort.
Blood test | third day
  Serum cortisol test (percentage of cortisol level in blood): It will take in the morning for two times one before the intervention or treatment in both groups and another one after 3 days to asses the pain level for patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: High power laser — https://doi.org/10.1016/j.jphotobiol.2017.05.022